CLINICAL TRIAL: NCT04635618
Title: A Pragmatic Superiority Randomized Controlled Trial Comparing Brief Cognitive Behavioral Telepsychotherapy, Brief Interpersonal Telepsychotherapy and Telepsychoeducation for the Reduction of Emotional Distress During COVID-19 Outbreak in Professionals and Students From Essential Services With a High Level of Emotional Distress in Brazil in the Context of COVID-19
Brief Title: Psychotherapy Strategies for the Treatment of Professionals and Students From Essential Services With High Levels of Emotional Distress in the Context of COVID-19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Principal Investigator, Giovanni Abrahao Salum Junior, Principal Investigator, Hospital de Clinicas de Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20200213_Treatment
Record Dates: First submitted 2020-11-05; First posted 2020-11-19 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Mental Disorder; COVID; Emotional Distress; Depression; Anxiety; Irritable Mood
MeSH Terms: conditions — Mental Disorders; Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Three-arm randomized clinical trial , including professionals and students from essential services suffering from high levels of anxiety, depression, and irritability symptoms during the COVID-19 outbreak randomized 1:1:1: to the Cognitive Behavioral Brief-Telepsychotherapy group (B-CBT, four sessions), Brief Interpersonal Telepsychotherapy (B-IPT, four sessions) or Telepsychoeducation group (a single session psychoeducation group plus weekly personalized pre-recorded videos for 4 weeks).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention I: Cognitive Behavioral Brief-Telepsychotherapy (Experimental): Four sessions of cognitive-behavioral therapy (CBT) conducted through a video call by a psychologist, accompanied by sending videos of 2 to 3 minutes with psychoeducational content and content related to CBT technique.
  Interventions: Behavioral: Cognitive Behavioral Brief-Telepsychotherapy
- Intervention II: Brief Interpersonal Telepsychotherapy (Experimental): Four sessions of interpersonal therapy (IPT) conducted by video call by a psychologist, accompanied by the sending of 2 to 3 minute videos with psychoeducational content and content related to the ITP technique.
  Interventions: Behavioral: Brief Interpersonal Telepsychotherapy
- Active Comparator: Telepsychoeducation group (Active Comparator): One single session of psychoeducation conducted through a video call by a psychologist, accompanied by sending videos of 2 to 3 minutes with psychoeducational content for 4 weeks.
  Interventions: Behavioral: Telepsychoeducation

INTERVENTIONS:
Behavioral: Cognitive Behavioral Brief-Telepsychotherapy — Four sections of Cognitive Behavioral Brief-Telepsychotherapy plus personalized pre-recorded videos
  Arms: Intervention I: Cognitive Behavioral Brief-Telepsychotherapy
Behavioral: Brief Interpersonal Telepsychotherapy — Four sections of Brief Interpersonal Telepsychotherapy plus personalized pre-recorded videos
  Arms: Intervention II: Brief Interpersonal Telepsychotherapy
Behavioral: Telepsychoeducation — A single session psychoeducation group plus weekly personalized pre-recorded videos for 4 weeks
  Arms: Active Comparator: Telepsychoeducation group

SUMMARY:
The study consists in a pragmatic superiority randomized controlled trial comparing different strategies of psychotherapy for professionals and students from essential services with high levels of emotional distress during the COVID-19 pandemic in Brazil. Therapeutic strategies to be evaluated are Brief Cognitive Behavioral Telepsychotherapy, Brief Interpersonal Telepsychotherapy and Telepsychoeducation, as an active control.

Note: This study was approved by the Ethics and Research Committee of the Hospital de Clínicas de Porto Alegre and is originally registered at Plataforma Brasil, a Brazilian study registration platform (under CAAE: 30608420.5.0000.5327). Recruitment began in May 28th 2020.

DETAILED DESCRIPTION:
PRAGMATIC TREATMENT TRIAL

TITLE: "A pragmatic superiority randomized controlled trial comparing Brief Cognitive Behavioral Telepsychotherapy, Brief Interpersonal Telepsychotherapy and Telepsychoeducation for the reduction of emotional distress during COVID-19 outbreak in professionals and students from essential services with a high level of emotional distress in Brazil".

IMPORTANCE: COVID-19 outbreak is associated with increased emotional distress (depression, anxiety, and irritability) all over the world. Currently, there are no large randomized trials testing interventions to reduce the burden caused by mental disorders during a pandemic outbreak of these proportions.

OBJECTIVE: To test the effectiveness of two modalities of Brief-Telepsychotherapy (Cognitive Behavioral and Interpersonal) to the reduction of symptoms of emotional distress (anxiety, depression, and irritability) in professionals and students from essential services with a high level of those symptoms in Brazil during the COVID-19 outbreak.

DESIGN, SETTING, AND PARTICIPANTS Thee-arm randomized clinical trial. Participants were recruited in Brazil from the national service of telehealth provided by the ministry of health. Participants included professional and students from essential services suffering from high levels of anxiety, depression, and irritability symptoms during the COVID-19 outbreak. High levels of symptoms were defined by either of the following: (1) T score higher than 70 on the PROMIS Anxiety Scale; (2) T score higher than 70 on the PROMIS Depression Scale; (3) T score higher than 70 on the PROMIS Anger Scale.

INTERVENTIONS: All participants will be randomized 1:1:1: to the Cognitive Behavioral Brief-Telepsychotherapy group (B-CBT, four sessions), Brief Interpersonal Telepsychotherapy (B-IPT, four sessions) or Telepsychoeducation group (a single session psychoeducation group plus weekly personalized pre-recorded videos for 4 weeks).

MAIN OUTCOMES AND MEASURES: The primary outcome will be the proportion of participants with a 50% reduction in T-scores in all the scales that were scored above 70 at baseline at 1-month. Secondary outcomes (1) the same measure of the primary outcome but measured at 3-month and 6-months follow-up; (2) mean score change in individual scales, quality of life and remission levels (proportion of patients with T-score of 50 or below in all of the four emotional distress subscales); (3) the same measure of the primary outcome but measured at midpoint (after the second session or 2-weeks); and (4) service satisfaction and net-promoter score at the end of the treatment.

EXPECTED RESULTS: To detect a 15% group difference between each group, an alpha of 0.017 (3 comparisons, 0,05/3), power of 90%, and 20% loss to follow up, we would need a total of 333 participants per group.

ELIGIBILITY:
Inclusion Criteria:

Professionals and students from essential services suffering from high levels of emotional distress

* T score higher than 70 on the PROMIS Anxiety Scale
* T score higher than 70 on the PROMIS Depression Scale
* T score higher than 70 on the PROMIS Anger Scale

Exclusion Criteria:

* Moderate to severe suicide risk assessed by a psychiatrist

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 999 (Estimated)
Dates: Start 2020-11-05 (Actual); Primary Completion 2021-07-13 (Estimated); Study Completion 2021-07-20 (Estimated)

PRIMARY OUTCOMES:
Symptom Reduction at 1-month | 1-month
  Proportion of participants with a 50% reduction in T-scores at 1-month in the scales Patient-Reported Outcomes Measurement Information System (PROMIS) of Depression, Anxiety and Anger that were scored above 70 at baseline.

SECONDARY OUTCOMES:
Symptom Reduction at 3 and 6-months follow-up | 3 and 6-month
  Proportion of participants with a 50% reduction in T-scores at 3 and 6-months follow-up in the scales Patient-Reported Outcomes Measurement Information System (PROMIS) of Depression, Anxiety and Anger that were scored above 70 at baseline measured
Remission Levels in distress scales | 1, 3 and 6-months
  Remission levels (proportion of patients with T-score of 50 or below) in distress scales (PROMIS of Depression, Anxiety and Anger)
Service Satisfaction | 1-month
  Service satisfaction measured by the net-promoter score at the end of the treatment (proportion of promoters - scores of 9 or 10)
Improvement in Quality of Life | 1, 3 and 6-months
  Mean score change in quality of life scale (PROMIS General Life Satisfaction Scale or GLSS)

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Salum, MD, PhD, Principal Investigator — Hospital de Clínicas de Porto Alegre, Porto Alegre/Brazil
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Plan to share study protocol, SAP, ICF, CRS, analytic code and individual-based variables.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Avaliable six months after study completion (antecipated - January 2022)
Access Criteria: Researchers and civil society

REFERENCES:
- [Derived] Damiano RF, Abreu M, Dreher CB, Bryan CJ, Miguel EC, Fleck M, Manfro GG, Salum GA. Risk Factors for Suicide Attempts and Psychiatric Hospitalization Among Brazilian Health Care Professionals. J Clin Psychiatry. 2025 Dec 31;87(1):25m15858. doi: 10.4088/JCP.25m15858. PMID 41499179
- [Derived] Martins DS, Viduani A, Dreher CB, Salum G, Manfro GG. Examining therapeutic alliance, adherence, and dropout in brief telepsychotherapy: A qualitative study. J Couns Psychol. 2025 Nov;72(6):699-709. doi: 10.1037/cou0000806. Epub 2025 Jun 2. PMID 40455512